CLINICAL TRIAL: NCT06128889
Title: Evaluation of a Supporting Transition and Resilience to Clinical Nursing Education (STRONG) Study - A Mixed Methods Evaluation
Brief Title: Evaluation of a Supporting Transition and Resilience to Clinical Nursing Education (STRONG) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NUS-IRB-2023-737
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Resilience; Practice Readiness; Depression; Anxiety; Stress; Physical Activity; Eating Behaviours
MeSH Terms: conditions — Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STRONG program (Experimental)
  Interventions: Behavioral: Supporting Transition and Resilience to Clinical Nursing Education (STRONG) Program

INTERVENTIONS:
Behavioral: Supporting Transition and Resilience to Clinical Nursing Education (STRONG) Program — The STRONG program adopts an asynchronous online learning approach and will be delivered over one week by a trained counsellor, and a nurse researcher. Students will attend an online self-paced program. The program will comprise of topics such as: (1) Resilience and protective factors, (2) introduction to clinical nursing education, (3) experiences of clinical attachments, and (4) stress, physical wellbeing and diet materials. Students will have access to online materials (e.g., short videos), have opportunities to discuss (e.g., forum) and infographics. Overall, the program will be delivered over in one week lasting six hours.

SUMMARY:
This study aims to address the following research questions:

1. Evaluate the effectiveness of a Supporting Transition and Resilience to Clinical Nursing Education (STRONG) program on first year nursing students' anxiety, depression, stress, resilience, practice readiness, physical activity and eating behaviours.
2. Explore first year nursing students' experiences and perception of the STRONG program.

Participants will be invited to participate in an asynchronous online STRONG program

ELIGIBILITY:
Inclusion Criteria:

* First year nursing students enrolled in the NUR1107B Nursing Practice Experience and NUR1202C Clinical Experience I module
* Above the ages of 18 years
* Able to comprehend the English language
* Have a device that can connect to the Internet

Exclusion Criteria:

* Students who refused to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Resilience | Before training
  Brief Resilience Scale
Resilience | Immediately after training
  Brief Resilience Scale
Resilience | 1 month after training
  Brief Resilience Scale
Depression, Anxiety, and Stress | Before training
  Depression, Anxiety and Stress Scale - 21
Depression, Anxiety, and Stress | Immediately after training
  Depression, Anxiety and Stress Scale - 21
Depression, Anxiety, and Stress | 1 month after training
  Depression, Anxiety and Stress Scale - 21
Practice Readiness | Before training
  Nursing Practice Readiness Scale
Practice Readiness | Immediately after training
  Nursing Practice Readiness Scale
Practice Readiness | 1 month after training
  Nursing Practice Readiness Scale
Physical activity | Before training
  International Physical Activity Questionnaire
Physical activity | Immediately after training
  International Physical Activity Questionnaire
Physical activity | 1 month after training
  International Physical Activity Questionnaire
Eating behaviours | Before training
  Self-regulation of Eating Behaviours Scale
Eating behaviours | Immediately after training
  Self-regulation of Eating Behaviours Scale
Eating behaviours | 1 month after training
  Self-regulation of Eating Behaviours Scale

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Ang, PhD, Principal Investigator — National University of Singapore

IPD SHARING:
Plan to Share IPD: Undecided